CLINICAL TRIAL: NCT07114718
Title: Starlight Cardiovascular Lifeline Ductus Arteriosus Stent IDE Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Starlight Cardiovascular Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G250132; 2R44HL158304-04A1 (NIH)
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Congenital Heart Disease; Congenital Heart Disease (CHD)
Keywords: Ductus Arteriosus Stent; pediatric stent; Lifeline Stent
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm - Treatment (Other): Treatment with the Lifeline Ductus Arteriosus Stent
  Interventions: Device: Ductus Arteriosus Stent

INTERVENTIONS:
Device: Ductus Arteriosus Stent — The eligible subjects will proceed to implantation of the Lifeline Ductus Arteriosus Stent to maintain patency of the PDA.
  Other Names: Stent; Pediatric Stent

SUMMARY:
Starlight Cardiovascular, Inc. is sponsoring a prospective, multi-center, study to evaluate safety and effectiveness of the Lifeline Ductus Arteriosus Stent System. The study device is a stent that is designed to maintain patency of the Ductus Arteriosus for children who need blood flow through that part of the heart.

DETAILED DESCRIPTION:
Starlight Cardiovascular, Inc. is sponsoring a prospective, multi-center, study to evaluate safety and effectiveness of the LifelineTM Ductus Arteriosus Stent System.

The purpose of the study is to determine whether the Ductus Arteriosus Stent System demonstrates safety and effectiveness for patients who require ductal patency and merits Food and Drug Administration (FDA) approval.

ELIGIBILITY:
Inclusion Criteria:

1. Parental or legal authorized representative provide consent for study enrollment
2. Infants < 6 months of age
3. Diagnosis of congenital heart defect with ductal-dependent pulmonary circulation requiring infusion of prostaglandins
4. Requires ductus arteriosus stent diameters of 3.5mm or 4mm and stent lengths between 16mm and 28mm

Exclusion Criteria:

1. Active blood stream infection
2. Active or history of endocarditis
3. Body weight <2.5kg
4. Gestational age <32 weeks at birth
5. Complete heart block
6. Total Anomalous Pulmonary Venous Return
7. Anatomic variation judged to be inappropriate for ductal stenting per the treating interventionalist
8. Presence of an aortopulmonary collateral that is expected to require unifocalization
9. Non-confluent pulmonary arteries (i.e. isolated pulmonary artery of ductal origin) or bilateral patent ductus arteriosus (PDA)
10. Pulmonary atresia with intact ventricular septum with RV-dependent coronary circulation
11. Currently participating in an investigational drug study or another device study that would confound the study results
12. Patient who is on extracorporeal membrane oxygenation (ECMO), ventricular assist device (VAD), or dialysis prior to ductal stenting procedure
13. Major co-morbidities which, in the opinion of the investigator, would negatively alter expected 1-year survival (e.g., intracranial hemorrhage, renal failure, etc.)
14. Patient who is undergoing another transcatheter procedure (e.g., atrial septostomy, aortic arch intervention, or right ventricular outflow tract intervention) during or within 24 hours prior to the ductus arteriosus stenting procedure
15. Patient who, at the time of enrollment, is deemed not to be a candidate for eventual stage II palliation of single ventricle heart disease, complete surgical repair, nor transcatheter treatment with resultant biventricular circulation
16. Patient who does not plan to return to the enrolling center or another participating center for stage II palliation, complete surgical repair, or definitive catheterization procedure
17. Contraindications to peri-procedural anticoagulation
18. Known to be non-responsive to aspirin or other antiplatelet therapies
19. Known hypersensitivity or allergy to Nickel
20. Known hypersensitivity to contrast media that cannot be adequately pre-medicated

Ages: 0 Minutes to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Implant to 30 days
  Freedom from death related to the device or implantation procedure or Major Complication related to the device or implantation procedure at 30 days.
Primary Efficacy Endpoint | Implant to 180 days
  Freedom from open surgical intervention to address stent dysfunction in subjects with a Lifeline stent implanted at the earlier of 180 days or the time of stent division or ligation during complete surgical repair or second stage surgery.

IPD SHARING:
Plan to Share IPD: No